CLINICAL TRIAL: NCT07309133
Title: Optimising Deep Brain Stimulation for Dystonia Using Local Field Potentials
Brief Title: Local Field Potentials in Dystonia
Acronym: LFP-DYT
Status: Recruiting | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Medtronic (Industry); Dystonia Europe (Unknown)
Responsible Party: Sponsor
Other Study IDs: 10878 - LFPDYT; 1982 (Other: Clinical Ageing Research Unit); 10878 (Other: Newcastle Hospitals R&D)
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Dystonia; Dystonia, Focal; Dystonia, Primary
Keywords: Deep Brain Stimulation; DBS; Globus Pallidus Interna; Local Field Potentials; Neurostimulation; Neurophysiology
MeSH Terms: conditions — Dystonia; Dystonic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cohort 1 (Pilot group): Description: First 3 participants with primary dystonia undergoing DBS. Used to optimize LFP sensing workflow and confirm the feasibility of data collection.
  Population: Adults (≥18 years) with primary dystonia scheduled for GPi DBS. Purpose: Workflow development and initial LFP data collection.
  Interventions: Device: Deep Brain Stimulation System
- Cohort 2 (Main observational group): Description: 8-10 participants with primary dystonia undergoing DBS and programmed using traditional clinical methods. LFP recordings are collected at each visit for correlation analysis.
  Population: Adults with primary dystonia (including idiopathic cervical dystonia and generalized dystonia).
  Purpose: Assess the relationship between LFP profiles and optimal stimulation sites determined by standard programming.
  Interventions: Device: Deep Brain Stimulation System
- Cohort 3 (Exploratory programming group): Description: 10-15 participants with primary dystonia who may receive programming guided by LFP analysis if interim results support feasibility.
  Population: Adults with primary dystonia undergoing DBS. Purpose: Explore whether LFP-guided programming improves clinical outcomes compared to traditional methods.
  Interventions: Device: Deep Brain Stimulation System

INTERVENTIONS:
Device: Deep Brain Stimulation System — The Medtronic Percept™ DBS system will be used as part of standard clinical care for dystonia. The study will utilize the device's sensing capabilities (BrainSense™) to record local field potentials for research purposes.

SUMMARY:
The goal of this clinical trial is to learn whether local field potential (LFP) signals recorded from the globus pallidus interna (GPi) using the Medtronic Percept™ deep brain stimulation (DBS) device can help optimize DBS programming for people with dystonia. The study will also explore whether LFP patterns can serve as a biomarker of disease activity and predict treatment response.

The main questions it aims to answer are:

Do LFP peaks in the alpha-theta range reliably correlate with dystonia severity and clinical characteristics? Can LFP-based programming achieve similar or better clinical outcomes compared to traditional programming methods? How do LFP profiles change with stimulation and other treatments such as botulinum toxin or oral medications?

Researchers will compare two programming approaches:

Traditional programming based on clinical assessment and imaging. LFP-guided programming based on the site and characteristics of LFP peaks

Participants will:

Undergo DBS surgery for dystonia as part of standard clinical care. Attend regular follow-up visits for DBS programming and outcome assessments. Complete clinical rating scales for dystonia severity, quality of life, cognition, and mood.

Take part in neurophysiological assessments, including surface EMG, EEG, and reaction time tasks.

Have LFP recordings collected using the Medtronic Percept™ device during clinic visits and, where possible, at home using device sensing features.

This study will help determine whether LFP analysis can shorten the time to optimal DBS settings and improve outcomes for people with dystonia.

DETAILED DESCRIPTION:
Dystonia is a disabling movement disorder characterized by sustained or intermittent muscle contractions that cause abnormal postures and movements. Deep brain stimulation (DBS) of the globus pallidus interna (GPi) is an established treatment for patients who do not respond adequately to first-line therapies such as botulinum toxin. However, clinical response to DBS in dystonia is highly variable, and optimization of stimulation settings often requires months of trial and error. This delay can prolong disability and increase healthcare burden.

Local field potentials (LFPs) are neural signals recorded from implanted DBS electrodes. In Parkinson's disease, LFP analysis has been used to guide programming and develop adaptive stimulation strategies. In dystonia, early studies suggest that low-frequency LFP peaks (typically in the alpha-theta range) may correlate with disease severity and optimal stimulation sites, but these findings have been limited to short-term recordings using externalized leads. The Medtronic Percept™ DBS system now allows chronic sensing of LFPs during routine clinical care, creating an opportunity to validate these observations and assess their clinical utility.

This single-site, prospective study will evaluate whether LFP profiles recorded from the GPi can guide DBS programming in patients with primary dystonia. The study includes an internal pilot phase followed by two main cohorts. Cohort 2 will undergo traditional programming based on clinical assessment and imaging, with LFP recordings collected at each visit. Cohort 3 will use an LFP-guided approach, selecting contacts and stimulation parameters based on the site and characteristics of LFP peaks. Participants will be followed for up to 12 months, with blinded video assessments and standardized rating scales to compare outcomes between programming strategies. Neurophysiological measures such as surface electromyography (EMG), electroencephalography (EEG), and reaction time tasks will also be collected to explore mechanistic links between stimulation and motor control.

The study aims to determine whether LFP analysis can shorten the time to optimal DBS settings and improve clinical outcomes compared to traditional methods. If successful, this approach could inform future development of adaptive DBS systems for dystonia, reducing variability in care and improving patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at screening.
* Clear clinical diagnosis of primary dystonia (idiopathic or genetic forms).
* Candidate for GPi DBS surgery for dystonia treatment.
* Able to provide informed consent.

Exclusion Criteria:

* Significant neurological or psychiatric disorder (including dementia) that would interfere with outcome evaluation.
* Participation in a therapeutic research trial within the last year.
* Diagnosis of functional (psychogenic) dystonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with a clinical diagnosis of primary dystonia (including idiopathic adult-onset focal cervical dystonia and young-onset generalized dystonia such as DYT1).
  All participants are scheduled to undergo deep brain stimulation (DBS) of the globus pallidus interna (GPi) as part of standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between GPi LFP peak characteristics and dystonia severity | Baseline (pre-activation) up to 1 year post-DBS activation
  Assess whether local field potential (LFP) peaks recorded from the globus pallidus interna using the Medtronic Percept™ DBS system correlate with clinical severity of dystonia as measured by standardized rating scales (e.g., TWSTRS for cervical dystonia, BFMDRS for generalized dystonia).

SECONDARY OUTCOMES:
Change in LFP peak amplitude with DBS stimulation | Activation visit and follow-up visits up to 12 months
  Assess whether DBS stimulation parameters reduce LFP peak amplitude in the alpha-theta range during programming sessions.
Relationship between LFP peak location and optimal stimulation contact | Baseline and follow-up to 12 months post-activation
  Evaluate whether the electrode contact with the highest LFP peak corresponds to the contact selected as optimal during traditional programming.
Association between LFP changes and clinical improvement | Baseline and follow-up until 12 months post-activation
  Investigate whether suppression or modulation of LFP peaks correlates with improvement in dystonia severity scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Ageing Research Unit,, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be stored securely and used only for approved analyses; summary results will be published.

REFERENCES:
- [Background] Ledingham D, Gibbs M, Mills R, Jenkins A, Nicholson C, Hussain MA, Baker M, Pavese N. Decoding Cervical Dystonia: Insights from Local Field Potentials in a Case Study Utilizing Open-Source Toolboxes. Mov Disord Clin Pract. 2025 Oct;12(10):1675-1678. doi: 10.1002/mdc3.70164. Epub 2025 Jun 5. No abstract available. PMID 40470846
- [Background] Ledingham D, Baker M, Pavese N. Local field potentials: Therapeutic implications for DBS in dystonia including adaptive DBS for dystonia. Deep Brain Stimulation. 2024;5:4-19. doi:10.1016/j.jdbs.2024.03.003